CLINICAL TRIAL: NCT01155973
Title: Educore Project: A Clinical Trial, Randomised by Clusters, to Assess the Effect of a Visual Learning Method on Blood Pressure Control in the Primary Health Care Setting
Brief Title: Educore Project: Effect of a Visual Learning Method for Improving Blood Pressure Control
Acronym: EDUCORE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gerencia de Atención Primaria, Madrid (Other Government)
Collaborators: Instituto de Salud Carlos III (Other Government); Fondo de Investigacion Sanitaria (Other)
Responsible Party: Principal Investigator, Esperanza Escortell, Epidemiologist, Gerencia de Atención Primaria, Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 09/90354
Record Dates: First submitted 2010-06-29; First posted 2010-07-02 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Hypertension
Keywords: Hypertension.; Cardiovascular risk.; Monitoring.; Primary health care.; Randomised controlled trial.; Cluster analysis
MeSH Terms: conditions — Hypertension | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EDUCORE intervention (Experimental): Use of low risk SCORE table. Use of visual impact images. Handing the patient a pamphlet (advice on how to maintain cardiovascular health plus the low risk SCORE table with the patient's current score marked).
  Interventions: Behavioral: EDUCORE intervention
- control group (Active Comparator): Use of low risk SCORE table; verbally informing the patient of his/her CVR. Giving advice/verbal information on risk factors.
  Interventions: Other: Control group

INTERVENTIONS:
Behavioral: EDUCORE intervention — Direct exhibition of their cardiovascular risk with SCORE, visual images and documentation to the patients
  Arms: EDUCORE intervention
Other: Control group — SCORE oral information and counseling as standard practice care
  Arms: control group

SUMMARY:
Background: High blood pressure (HBP) is a major risk factor for cardiovascular disease (CVD). European hypertension and cardiology societies as well as expert committees on CVD prevention recommend stratifying cardiovascular risk (CVR) using the SCORE method, the modification of lifestyles to prevent CVD, and achieving good control over risk factors. The EDUCORE (Education and Coronary Risk Evaluation) project aims to determine whether the use of a CVR visual learning method - the EDUCORE method - is more effective than normal clinical practice in improving the control of blood pressure within one year in patients with poorly controlled hypertension but no background of CVD.

Design & Method: Cluster randomized controlled clinical trial. Location: 22 primary health care centres in Madrid. Participants: patients diagnosed as hypertensive (systolic >140 mmHg and/or diastolic >90 mmHg) at least a year before, uncontrolled. Age: 40-65 year-old patients who consent to take part. Sampling: randomized cluster assignment. Random allocation unit: health care centre. Analysis unit: patient who match criteria. Size: 736 patients (368 each arm. Measurements: Outcome variables: systolic and diastolic blood pressure (mmHg). Cardiovascular risk level: SCORE. Measure of Adherence to treatment (Morisky-Green questionnaire. Health related quality of life questionnaire MINICHAL. Smoking habits. Total Cholesterol. Other variables: Gender. Age. Educational level. Physical activity in metabolic equivalent (MET). Body mass index. Drug consume (cardiovascular line). Treatment changes and nature of the change. Intervention: EDUCORE group (direct exhibition of their cardiovascular risk with SCORE, visual images and documentation to the patients); Control Group: standard practice care.

DETAILED DESCRIPTION:
Aim: To measure the effectiveness of an educational intervention in uncontrolled hypertensive patients without cardiovascular disease (primary prevention), compared with clinical practice to improve hypertension control in a year.

Method: This work describes a protocol for a clinical trial, randomised by clusters and involving 22 primary healthcare clinics (PHCC), to test the effectiveness of the EDUCORE method. The number of patients required was 736, all between 40 and 65 years of age (n=368 in the EDUCORE and control groups), all of whom had been diagnosed with HBP at least one year ago, and all of whom had poorly controlled hypertension (systolic blood pressure ≥ 140 mmHg and/or diastolic ≥ 90 mmHg). All personnel taking part were explained the trial and trained in its methodology. The EDUCORE method contemplates the visualisation of low risk SCORE scores using images embodying different stages of a high risk action, plus the receipt of a pamphlet explaining how to better maintain cardiac health. The main outcome variable was the control of blood pressure; secondary outcome variables included the SCORE score, therapeutic compliance, quality of life, and total cholesterol level. All outcome variables were measured at the beginning of the experimental period and again at 6 and 12 months. Information on sex, age, educational level, physical activity, body mass index, consumption of medications, change of treatment and blood analysis results was also recorded.

Information source: Clinical interview and assessments tests. The data will be registered in Electronic data capture system.

Statistical Analysis: Primary and secondary effectiveness. Adjusting by prognosis factors with random effects models (logistic regression) (dependent variable: good/bad blood pressure control; independent variable: intervention group).

Discussion: The EDUCORE method could provide a simple, inexpensive means of improving blood pressure control, and perhaps other health problems, in the primary healthcare setting.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed as hypertensive (systolic >140 mmHg and/or diastolic >90 mmHg) at least a year before, uncontrolled.
* Age: 40-65 year-old patients
* Patients who consent to take part

Exclusion Criteria:

* Diabetes Mellitus
* Cardiovascular disease...

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 452 (Actual)
Dates: Start 2010-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Main outcome variable: control of blood pressure | Baseline and 1 year
  Blood pressure (bp): systolic and diastolic blood pressure, determined using the Riva-Rocci method and listening for Korotkoff sounds, using validated and calibrated sphygmomanometers. Control BP: SBP < 140 mmHg and DBP < 90 mmHg

SECONDARY OUTCOMES:
Cardiovascular risk (CVR) level : Use of low risk SCORE table | Baseline and 1 year
  Calculation of CVR at appointments 1, 3 and 5 (at the beginning of the experimental period and again at 6 and 12 months).
  Calculation of the projected CVR at 60 years of age for all patients under this age.
Measure of Adherence to treatment (Morisky-Green questionnaire) | 1 year
  therapeutic compliance (measured using the Morisky-Green treatment compliance questionnaire)
Smoking habits | Baseline and 1 year
  Use of tobacco
Total Cholesterol | Baseline and 1 year
  Total cholesterol level

CONTACTS AND LOCATIONS:
Overall Officials: Esperanza Escortell, MD, Principal Investigator — Gerencia de Atención Primaria, Madrid
Locations (1):
- Gerencia de Atención Primaria, Madrid, Madrid, Spain

REFERENCES:
- [Background] Rodriguez-Salceda I, Escortell-Mayor E, Rico-Blazquez M, Riesgo-Fuertes R, Asunsolo-del Barco A, Valdivia-Perez A, del Cura-Gonzalez I, Garcia-Canon AB, Ortiz-Jimenez MF, Cabello-Ballesteros L, Garrido-Elustondo S, Chamorro-Gonzalez L, Rodriguez-Barrientos R; EDUCORE Group. EDUCORE project: a clinical trial, randomised by clusters, to assess the effect of a visual learning method on blood pressure control in the primary healthcare setting. BMC Public Health. 2010 Jul 30;10:449. doi: 10.1186/1471-2458-10-449. PMID 20673325
- [Derived] Lindson N, Pritchard G, Hong B, Fanshawe TR, Pipe A, Papadakis S. Strategies to improve smoking cessation rates in primary care. Cochrane Database Syst Rev. 2021 Sep 6;9(9):CD011556. doi: 10.1002/14651858.CD011556.pub2. PMID 34693994